CLINICAL TRIAL: NCT01455051
Title: Ofatumumab as Part of the Reduced Intensity Conditioning Regimen for Patients With High Risk Chronic Lymphocytic Leukemia Undergoing Allogeneic Hematopoietic Cell Transplantation: a Pilot Study by GETH and GELLC
Brief Title: Ofatumumab as Part of Reduced Intensity Conditioning (RIC) Regimen for Patients With High Risk Chronic Lymphocytic Leukemia (CLL) Undergoing Allogeneic Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETH-CLL4; 2010-024467-40 (EudraCT Number)
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): We plan to add five doses of ofatumumab to the standard conditioning regimen (fludarabine + melphalan). Ofatumumab will be administered on days -20 (300 mg), -13 (2000 mg), -6 (2000 mg), +1 (1000 mg) and +8 (1000 mg) of the transplantation (day 0 being the day of the hematopoietic cell infusion). If the patient requires donor lymphocyte infusions within 3 years after the procedure, these infusions will also include one administration of 300 mg of ofatumumab, followed by a 1000 mg dose, 7 days later).
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — We plan to add five doses of ofatumumab to the standard conditioning regimen (fludarabine + melphalan). Ofatumumab will be administered on days -20 (300 mg), -13 (2000 mg), -6 (2000 mg), +1 (1000 mg) and +8 (1000 mg) of the transplantation (day 0 being the day of the hematopoietic cell infusion). If the patient requires donor lymphocyte infusions within 3 years after the procedure, these infusions will also include one administration of 300 mg of ofatumumab, followed by a 1000 mg dose, 7 days later).
  Other Names: Arzerra

SUMMARY:
A good proportion of patients with chronic lymphocytic leukemia (CLL) can be managed effectively with palliative chemotherapy. However, there is a group of younger patients with poor risk disease whose life expectancy is significantly reduced. As a result, reduced intensity conditioning (RIC) allogeneic hematopoietic cell transplantation (allo-HCT) has been investigated as a potentially curative procedure.

Recently, the European Group for Blood and Marrow Transplantation (EBMT) published a set of guidelines suggesting situations where allo-HCT might be considered a therapeutic option for CLL patients. Their conclusions were that allo-HCT was reasonable for younger CLL patients refractory to fludarabine, relapsing within two years of intensive treatment, or with p53 abnormalities requiring treatment.

However, the results with RIC allo-HCT are not entirely satisfactory, and progression-free survival after allo-HCT revolves around 35-40% at 3-5 years following allo-HCT. This is due to non-relapse mortality, which is significantly associated with the development of graft-versus-host disease (GVHD), but also due to disease relapse. These relapses may occur early in the course of the transplantation, like any other hematological malignancy, but late relapses have also been reported.

Several strategies have been tested in order to improve these results. The anti-CD20 monoclonal antibody rituximab, given concomitantly with allo-HCT or donor lymphocyte infusions, may reduce graft-versus-host disease and facilitate disease control. This may be due, not only to direct cytotoxicity, but also to modulation of GVHD and the graft-versus CLL effect (GVCLL). Interestingly, rituximab has been shown to promote the cross-presentation of tumor-derived peptides by antigen-presenting cells, thus enhancing the formation of cytotoxic T-cell clones and a GVCLL effect. With the addition of rituximab to the conditioning regimen, rates at 4 years for current progression-free survival (CPFS) and overall survival were 44% and 48%.

The investigators hypothesize that ofatumumab, having a more potent anti-CLL activity and complement-dependent cytoxicity than rituximab, could improve disease control and modulate the GVCLL effect more effectively, thus reducing the GVHD rate and subsequently improving the non-relapse mortality and progression-free survival in the long term.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with CD20+ chronic lymphocytic leukemia according to the World Health Organization.
2. Patients older than 18 and younger than 70 years old.
3. Patients who failed to meet NCI Working Group criteria for complete or partial response after therapy with regimens containing fludarabine or with disease relapse within 12 months after completing therapy with fludarabine containing regimen. Patients not eligible for fludarabine treatment, could also be included provided the disease remains unresponsive or relapses with 12 months after completing alternative salvage regimens (i.e. autologous HCT, bendamustine, gemcitabine, alemtuzumab or high-dose methyl-prednisolone), OR Patients with novo or acquired "17p deletion" cytogenetic abnormality. These patients must have received induction chemotherapy but could be transplanted in first complete or partial response.
4. Patients must have achieved a complete or partial response after the last therapy given prior to transplantation. Patients with clinically suspected or histologically confirmed Richter's transformation could be included if they are in complete response at the time of transplantation.
5. Patients who have not received more than four lines of therapy prior to transplantation.
6. Patients who have suitable HLA-matched related or unrelated donors willing to receive G-CSF, undergo apheresis to collect PBMC, and to donate stem cells. Patients with a single-locus mismatched donor available are also eligible.
7. ECOG functional status of 0 to 2.
8. Life expectancy of at least 6 months.
9. Signed informed consent.

Exclusion Criteria:

* Intolerance to rituximab or any other anti-CD20 monoclonal antibody.
* Diagnosis of CNS involvement with CLL.
* Prior allogeneic HCT.
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Active infection unresponsive to medical therapy such as, but not limited to, chronic renal infection, chronic chest infection, tuberculosis and active hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
* Known HIV positive.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result.
* Severe organ dysfunction as defined by: cardiac ejection fraction <40%; DLCO <40%; calculated GFR < 30 ml/min; or bilirubin > 3 times the upper normal limit (unless due to CLL or Gilbert syndrome).
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
CPFS at 3y | At 3 years
  Current progression-free survival (CPFS) at 3 years.

SECONDARY OUTCOMES:
CPFS at 5y | At 5 years
  Current progression-free survival (CPFS) at 5 years
NRM at 1/5 years | At 1 and 5 years
  Non-relapse mortality at 1 and 5 years
Acute GVHD at 3mo | At 3 months
  Incidence of acute graft-versus-host disease, grade II-IV, at 3 months
Chronic GVHD at 1/5y | At 1 and 5 years
  Incidence of extensive chronic graft-versus-host disease at 1 and 5 years
Toxicity criteria | During all 3 years
  Evaluation of toxicity following common toxicity criteria, release 3.0
OS at 3/5y | At 3 and 5 years
  Overall survival at 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Julio Delgado, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (9):
- Spain (9):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat
  - Hospital La Princesa, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Clinico, Valencia
  - Hospital La Fe, Valencia

REFERENCES:
- [Result] Montesinos P, Cabrero M, Valcarcel D, Rovira M, Garcia-Marco JA, Loscertales J, Moreno C, Duarte R, Terol MJ, Villamor N, Abrisqueta P, Caballero D, Sanz J, Delgado J. The addition of ofatumumab to the conditioning regimen does not improve the outcome of patients with high-risk CLL undergoing reduced intensity allogeneic haematopoietic cell transplantation: a pilot trial from the GETH and GELLC (CLL4 trial). Bone Marrow Transplant. 2016 Oct;51(10):1404-1407. doi: 10.1038/bmt.2016.145. Epub 2016 May 23. No abstract available. PMID 27214073
- See also: Related Info — http://www.nature.com/bmt/journal/vaop/ncurrent/full/bmt2016145a.html